CLINICAL TRIAL: NCT06655207
Title: Pivotal, Prospective, Multi-centre, Single-arm Study to Evaluate the Safety and Effectiveness of Oli for Identification of Patients, During the Intrapartum Period, Who Are at Higher Risk of Developing Abnormal Postpartum Uterine Bleeding, Including Postpartum Haemorrhage, in Advance of Delivery/Birth
Brief Title: Pivotal, Prospective, Multi-centre, Single-arm Study to Evaluate the Safety and Effectiveness of Oli for Identification of Patients, During the Intrapartum Period, Who Are at Higher Risk of Developing Abnormal Postpartum Uterine Bleeding, Including Postpartum Haemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baymatob Operations Pty Ltd (Industry)
Collaborators: Royal North Shore Hospital (Other); Royal Hospital For Women (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OLIPPH-CI-2201
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Post Partum Haemorrhage; Maternal Care Patterns; High Risk Pregnancy
Keywords: Pivotal Study; Single arm; prospective
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Oli is a non-invasive, wearable device, designed to provide clinicians with an early indication if the participant is at a higher risk of developing abnormal postpartum uterine bleeding — Oli is a non-invasive wearable device, designed to provide clinicians with an early indication if the participant is at a higher risk of developing abnormal postpartum uterine bleeding, including postpartum haemorrhage.

SUMMARY:
Oli is a predictive, non-invasive device, intended to be placed on the participant's maternal abdomen during the intrapartum period, which can alert healthcare professionals of an impending cumulative blood loss of ≥500 ml (abnormal postpartum uterine bleeding) or cumulative blood loss of ≥1000ml (postpartum haemorrhage) at least 1 hour in advance of birth. This study is being undertaken to assess the performance of Oli measuring cumulative blood loss ≥500ml and ≥1000ml, as well as evaluate its safety profile.

DETAILED DESCRIPTION:
The World Health Organization (WHO) recognizes postpartum haemorrhage as a blood loss of 500ml or more within 24 hours after delivery and severe PPH as a blood loss of 1000ml within the same timeframe [2]. The American College of Obstetricians and Gynaecologists (ACOG) defines PPH as a cumulative blood loss of greater than or equal to 1000ml or blood loss accompanied by signs and symptoms of hypovolemia within 24 hours after the birth process [7] and recognizes a blood loss greater than 500ml as abnormal, and should be treated as a Stage 1 Obstetric Haemorrhage [17]. Further, the CMQCC Obstetric Haemorrhage Care Guidelines identifies a blood loss greater than 500ml as the trigger for the activation of haemorrhage protocols [18]. The Royal Australin and New Zealand College of Obstetricians and Gynaecologists (RANZCOG) also recognises postpartum haemorrhage as a blood loss of 500ml or more within 24 hours after delivery [26]. Consistent with these standards, Baymatob for the purpose of this study has defined Abnormal Postpartum Uterine Bleeding as postpartum blood loss ≥ 500ml.

Oli is a non-invasive device that uses several different parameters to identify those individuals who are likely to experience an APUB, including PPH, prior to birth. Oli has been granted FDA Breakthrough Device Designation for use by healthcare providers to identify a patient, during the intrapartum period, who is at higher risk of developing abnormal postpartum uterine bleeding, including postpartum haemorrhage, in advance of delivery/birth.

Oli functions by capturing physiological signals (a combination of biopotentials, skin temperature, movement and deformation of the maternal abdomen) via a wearable sensor attached to the maternal abdomen by electrodes during the intrapartum period. The physiological signals are processed and analysed via a fixed machine learning algorithm against a pre-defined threshold that indicates whether an individual is at an increased risk of APUB including PPH occurring.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Provision of informed consent i.e. participant must be able to understand and sign the Participant Information and Consent Form
* ≥28 weeks gestation
* Planning for normal vaginal delivery (participants requiring emergency caesarean delivery will not be excluded)

Exclusion Criteria:

* Currently participating in an investigational study that in the Investigator's opinion makes it undesirable to participate in this trial.
* Known significant sensitive skin or allergy/hypersensitivity to the medical gel/adhesive used to adhere the electrodes to the body
* Any concurrent condition which in the Investigator's opinion makes it undesirable for the participant to participate in the trial or which would jeopardize compliance with the protocol or follow up.
* Participant was monitored in the intrapartum period in the Oli Pilot Study (ETH00410).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Assess the performance of Oli as calculated by comparing the output of Oli (up to 1 hour prior to birth) against the clinically documented value of cumulative blood loss ≥ 500ml or any blood loss with signs and/or symptoms of hypovolemia within 24 hour | 6 months
To assess the performance of Oli in cumulative blood loss ≥ 1000ml (ACOG) | 14 months

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - UC Health University of Colorado Hospital, Denver, Colorado
  - Woman's Hospital, Baton Rouge, Louisiana
  - Columbia University Irving Medical Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - UPMC Magee Womens Hospital, Pittsburgh, Pennsylvania
- Australia (2):
  - Royal Hospital for Women, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales

IPD SHARING:
Plan to Share IPD: Undecided